CLINICAL TRIAL: NCT01314222
Title: A Randomized, Multicenter, Double-blind, Placebo and Active-controlled, Cross-over Study of the Efficacy and Safety of BMS-954561 in Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Brief Title: Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CN169-001; 2010-023042-70 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-03-14 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: BMS-954561 40mg or 80mg (Other): BMS-954561 40mg or 80mg TID to Placebo OR Placebo to 40mg or 80mg TID
  Active to Placebo or Placebo to Active (cross-over)
  Interventions: Drug: BMS-954561; Drug: Placebo matching BMS-954561
- Arm 2: BMS-954561 150mg or 300mg (Other): BMS-954561 150mg or 300mg TID to Placebo OR Placebo to 150mg or 300mg TID
  Active to Placebo or Placebo to Active (cross-over)
  Interventions: Drug: BMS-954561; Drug: Placebo matching BMS-954561
- Arm 3: Pregabalin 100mg (Other): Pregabalin 100mg TID to Placebo OR Placebo to 100mg TID
  Active to Placebo or Placebo to Active (cross-over)
  Interventions: Drug: Pregabalin; Drug: Placebo matching Pregabalin

INTERVENTIONS:
Drug: BMS-954561
  Arms: Arm 1: BMS-954561 40mg or 80mg; Arm 2: BMS-954561 150mg or 300mg
Drug: Pregabalin
  Arms: Arm 3: Pregabalin 100mg
Drug: Placebo matching BMS-954561
  Arms: Arm 1: BMS-954561 40mg or 80mg; Arm 2: BMS-954561 150mg or 300mg
Drug: Placebo matching Pregabalin
  Arms: Arm 3: Pregabalin 100mg

SUMMARY:
The purpose of the study is to evaluate the efficacy of study drug (BMS-954561) as compared to placebo in the treatment of patients with diabetic peripheral neuropathic pain (DPNP).

DETAILED DESCRIPTION:
Allocation: Randomized Stratified; Intervention Model: Cross-over Versus Comparator + Placebo

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetes with painful, distal, symmetrical, sensory-motor neuropathy attributed to diabetes, of at least 6 months duration.
* Score of ≥3 on Michigan Neuropathy Screening Instrument
* The patient is able to satisfactorily complete, in the Investigator's judgment, the Cognitive Battery.
* Based on patient diary information collected during the Screening/Baseline period, the patient has completed at least 5 of 7 daily diary entries and has an average weekly pain rating of at least 4 on the 11-point pain rating scale, in the week immediately prior to randomization (Baseline Visit).
* Male or female, 18-85 years of age.

Exclusion Criteria:

* History of complete lack of response to Pregabalin (at least 300 mg qd for 4 weeks) or Gabapentin (at least 1800 mg qd for 4 weeks).
* Other severe pain that may potentially confound pain assessment.
* Hemoglobin A1c > 9%
* Hemoglobin ≤ 9 g/dL
* Estimated glomerular filtration rate (eGFR) according to the re-expressed abbreviated (four-variable) Modification of Diet in Renal Disease (MDRD) Study equation ≤ 50ml/min/1.73m2
* Patients who have been on a stable dose of anticonvulsant, anticholinergic, diabetic meds, nicotine replacements, or any other smoking cessation meds for <4 weeks prior to randomization. Patients who are on stable doses for ≥ 4 weeks prior to randomization are allowed, however, there should be no adjustments to the dose of these medications during study.
* Patients currently on more than one drug for treatment of neuropathic pain (low dose opioids or antidepressants). Patients are allowed to participate if on a stable dose of for at least 4 weeks prior to randomization (Day1) and should remain stable during study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the average pain score for BMS-954561 vs. placebo. | Up to 10 weeks

SECONDARY OUTCOMES:
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Screening/Baseline Phase: Baseline
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 1
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 2
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 3
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 4
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 5
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 6
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 7
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 8
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 9
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Double-blind Treatment Phase: Week 10
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 2
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 4
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 8
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 12
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 16
Evaluate the effect of BMS-954561 compared to placebo using the Brief Pain Inventory-short form (BPI-SF). | Open-Label Phase: Week 20
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 1
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 2
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 3
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 4
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 5
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 6
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 7
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 8
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 9
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Double-blind Treatment Phase: Week 10
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 2
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 4
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 8
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 12
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 16
Evaluate the effect of BMS-954561 compared to placebo, on the Patient Global Impression of Change (PGIC) scale. | Open-Label Phase: Week 20
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Screening/Baseline Phase: Baseline
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 1
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 2
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 3
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 4
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 5
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 6
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 7
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 8
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 9
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Double-blind Treatment Phase: Week 10
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 2
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 4
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 8
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 12
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 16
Evaluate the tolerability and safety of BMS-954561 in patients with DPNP as measured by the frequency and severity of adverse events, frequency of severe adverse events, and discontinuations due to adverse events. | Open-Label Phase: Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (21):
  - Achieve Clinical Research, Llc, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Torrance Clinical Research, Lomita, California
  - Office Of Richard S. Cherlin, Md, Los Gatos, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Brain Matters Research, Delray Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Llc, Orlando, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Northwest Neurology Ltd., Lake Barrington, Illinois
  - Commonwealth Biomedical Research, Llc, Madisonville, Kentucky
  - The Center For Pharmaceutical Research. Pc, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Finger Lakes Clinical Research, Rochester, New York
  - Physicians East P.A., Greenville, North Carolina
  - Pmg Research Of Winston-Salem, Winston-Salem, North Carolina
  - Radiant Research, Inc., Akron, Ohio
  - Neurology & Neuroscience Center Of Ohio, Toledo, Ohio
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
- France (3):
  - Local Institution, Dijon
  - Local Institution, Nantes
  - Local Institution, Nice

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx